CLINICAL TRIAL: NCT04065997
Title: Apogee International
Status: Terminated | Type: Observational
Why Stopped: Due to Medtronic's decisions to stop sales and distribution of the HVAD System and subsequent stop of study enrollments, limited data will be available. Therefore it is not expected to provide new insights.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Apogee International
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients implanted with HVAD System: Patients intended to be implanted with a HeartWare HVAD per the current (local) guidelines, are eligible for enrollment into Apogee International and must be consented for Apogee International prior to the HVAD implant.
  Interventions: Device: HeartWare Ventricular Assist Device

INTERVENTIONS:
Device: HeartWare Ventricular Assist Device — The HVAD is an implantable centrifugal rotary blood pump that is implanted in the pericardial space and is designed to provide up to 10 L/min of blood flow from the left ventricular to the aorta. The HVAD System is comprised of three major components: the HVAD (pump) with inflow and outflow conduits, a Controller (microprocessor unit that controls the operation of the HVAD), and power sources (AC and DC power adapters that provide power to the Controller and implanted HVAD).
  Other Names: HVAD

SUMMARY:
Medtronic is sponsoring the Apogee International registry to further confirm safety and efficacy of the HVAD™ System when used as intended, in "real world" clinical practice and to enhance scientific understanding of the implant procedure, optimized blood pressure management, anticoagulation/ antiplatelet therapies, logfile analysis and acoustic spectrum analysis in patients receiving a Medtronic HeartWare™ HVAD™ for bridge to transplant and destination therapy indications.

DETAILED DESCRIPTION:
Apogee International is a prospective, non-interventional, post-market, multi-site registry, conducted within Medtronic's Product Surveillance Registry (PSR) Platform. Enrollment into Apogee International will be comprised of newly implanted, commercial use patients with the HeartWare Ventricular Assist Device System (HVAD System).

Sites selected to participate are expected to collect data in at least one of these five modules:

1. Logfile Download;
2. Anti-coagulation / Anti-platelet Management;
3. Blood Pressure (BP) Management;
4. Acoustic Spectrum Analysis;
5. Infection Control

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements;
* Enrollment into Apogee International will be comprised of newly enrolled, commercial use patients with the HeartWare HVAD System;
* Patient is consented prior to the HVAD implant procedure.

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up;
* Participation is excluded by local law;
* Patient is currently enrolled or plans to enroll in concurrent drug/device study that may confound the PSR results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients intended to be implanted with a HeartWare HVAD per the current (local) guidelines, are eligible for enrollment into Apogee International and must be consented for Apogee International prior to the HVAD implant.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Major adverse events | Implant to 12 months
  Major adverse events are defined to be occurrence of major infection, major bleeding, device malfunction, stroke or death.

CONTACTS AND LOCATIONS:
Locations (31):
- St. Vincents Hospital, Sydney, Australia
- Medical University of Vienna, Vienna, Austria
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium
- Aarhus Universitetshospital, Aarhus, Denmark
- Helsinki University Hospital, Helsinki, Finland
- Germany (9):
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bad Oeynhausen
  - Schuechtermann Klinik, Bad Rothenfelde
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Herzzentrum Leipzig GmbH, Leipzig
  - Otto von Guericke Universitat - Universitätsklinikum Magdeburg, Magdeburg
  - Eberhard Karls Universität Tübingen - Universitätsklinikum Tübingen, Tübingen
- Italy (3):
  - Azienda Ospedaliero Universitaria S. Orsola Malpighi Bologna, Bologna
  - Ospedale San Raffaele, Milan
  - ISMETT, Palermo
- National Research Cardiac Surgery Center, Astana, Kazakhstan
- Al Rassoul Al Azam Hospital - Beirut Cardiac Institute, Beirut, Lebanon
- Netherlands (2):
  - Leiden Universitair Medisch Centrum (LUMC), Leiden
  - University Medical Center Utrecht, Utrecht
- Oslo Universitetssykehus-Rikshospitalet, Oslo, Norway
- Instytut Kardiologii, Warsaw, Poland
- Klinicki Centar Srbije, Belgrade, Serbia
- Spain (2):
  - Hospital Universitario da Coruña, A Coruña
  - Hospital Universitari de Bellvitge, Barcelona
- UniversitätsSpital Zürich, Zurich, Switzerland
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Ankara
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
- United Kingdom (2):
  - Royal Brompton & Harefield NHS Foundation Trust - Harefield Hospital, Harefield
  - Freeman Hospital, Newcastle